CLINICAL TRIAL: NCT05442138
Title: A Prospective Observational Study on the Potential Benefit of Neoadjuvant Therapy for Advanced Gastric Cancer Based on Organoid Drug Susceptibility Screening
Brief Title: A Study on the Potential Benefit of Neoadjuvant Therapy for AGC Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: OneTar
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-06

CONDITIONS: Early Gastric Cancer; Tumor Organoids
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Early gastric cancer（AGC）has no effective characteristic symptoms and signs according to clinical statistics. Neoadjuvant chemotherapy (NAC) significantly reduces the size of AGC tumors so that it has become the recommended treatment for AGC in major guidelines. However, Some patients miss the best time for surgical treatment and may have irreversible chemotherapy side effects due to NAC lacks the guidance of new indicators for precise treatment such as molecular biomarkers. Tumor organoids are highly consistent with the clinical drug sensitivities of patients which could be used as clinical treatment prediction models thus providing guidance for individualized medicine. Therefore, the project is the first to carry out the prospective study by screening the potential benefit populations of NAC based on tumor organoids drug susceptibility experiment. The following hypothesis are put forward：the potential benefit population of NAC screened by tumor organoid drugs susceptibility technology will have better clinical efficacy, better treatment tolerance and higher adverse reaction rate.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75 years old;
2. Qualitative diagnosis: gastroscopic biopsy confirmed adenocarcinoma;
3. Localization diagnosis: the tumor is located in the stomach or gastroesophageal junction;
4. The clinical staging is stage III:

   A. Assess tumor stage: T3-4N1-2; B. Excluding distant organ metastasis (M0);
5. Physical condition (ECOG) score ≤ 1 point;
6. Those with effective preoperative neoadjuvant therapy and successful surgery agreed to receive 5 cycles of standard SOX chemotherapy after surgery;
7. Sign the informed consent form and be willing to participate in this project.

Exclusion Criteria:

1. Simultaneous or metachronous multiple primary malignant tumors;
2. Preoperative imaging examination results showed that there was distant metastasis;
3. Preoperative imaging findings:

   A. The tumor involving surrounding organs requires combined organ resection; B. Distant organ metastases; C. Those who cannot perform R0 resection;
4. Past history of malignant tumor;
5. Abnormal heart, lung, liver, kidney, hematopoietic function and bone marrow reserve function, unable to tolerate surgical treatment and chemotherapy;
6. Mental illness or other serious cardiovascular disease;
7. Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with AGC who need NAC before radical surgery.
Sampling Method: Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | time before the surgery
Tumor Regression Grading | time before the surgery